CLINICAL TRIAL: NCT02285257
Title: Epidemiology of Sepsis at Yuetan Subdistrict in Beijing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MICU2014-1; Z131107002213112 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Sepsis
Keywords: Sepsis, Severe sepsis, septic shock, epidemiology, outcome
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the epidemiology and outcome of sepsis at Yuetan subdistrict in Beijing in mainland China).

DETAILED DESCRIPTION:
1. Questionnaires were used to collect the characteristic information of people living in Yuetan subdistrict in Beijing and select people who had been hospitalized because of any reasons between July 2012 and June 2014.
2. Data were collected on all patients admitted into different hospitals during the study period. The following information was recorded:demographic characteristics and admission category (whether medical, scheduled surgery, nonoperative trauma, or unscheduled surgery), presence of preexisting organ insufficiency,using definitions included in the Acute Physiology and Chronic Health Evaluation (APACHE) II score11; co- morbidities and the estimated prognosis of any preexisting underlying disease, following the classification of McCabe and Jackson.
3. Patients were included in the study cohort when having, in association with a documented or strongly suspected infection and fullfil the diagnostic criteria of sepsis according to the "Surviving Sepsis Campaign: International guidelines for management of severe sepsis and septic shock:2012".

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Having lived in Yuetan Subdistirct for at least 1 year
* Having, in association with a documented or strongly suspected infection and fullfil the diagnostic criteria of sepsis according to the "Surviving Sepsis Campaign:International guidelines for management of severe sepsis and septic shock:2012"

Exclusion Criteria:

* Age<18 years
* Lived in Yuetan Subdistrict less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Questionnaires were used to collect the characteristic information of people living in Yuetan subdistrict in Beijing for more than 1 years people who had been hospitalized because of any reasons between July 2012 and June 2014 were selected.Patients were included in the study cohort when having, in association with a documented or strongly suspected infection and fullfil the diagnostic criteria of sepsis according to the "Surviving Sepsis Campaign:International guidelines for management of severe sepsis and septic shock:2012".
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
incidence of sepsis of people living in Yuetan subdistrict in Beijing | 2012-7-1~2014-6-30, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, professor, Study Director — Medical ICU, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences
Locations (1):
- MICU of Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian HC, Zhou JF, Weng L, Hu XY, Peng JM, Wang CY, Jiang W, Du XP, Xi XM, An YZ, Duan ML, Du B; for China Critical Care Clinical Trials Group (CCCCTG). Epidemiology of Sepsis-3 in a sub-district of Beijing: secondary analysis of a population-based database. Chin Med J (Engl). 2019 Sep 5;132(17):2039-2045. doi: 10.1097/CM9.0000000000000392. PMID 31425273